CLINICAL TRIAL: NCT02494336
Title: Trans-incisional Rectus Sheath Block Versus Laparoscopic Guided Rectus Sheath Block for Pediatric Single Incision Laparoscopic Cholecystectomy: A Prospective, Randomized Study
Brief Title: Trans-incisional vs Laparoscopic Guided Rectus Sheath Block for Pediatric Single Incision Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00041111
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trans-incisional rectus sheath block (Active Comparator): rectus sheath block under direct visualization through the umbilical incision by the attending surgeon
  Interventions: Procedure: Trans-incisional rectus sheath block; Drug: Ropivacaine
- Laparoscopic guided rectus sheath block (Active Comparator): rectus sheath block under direct laparoscopic visualization by the attending surgeon
  Interventions: Procedure: Laparoscopic guided rectus sheath block; Drug: Ropivacaine

INTERVENTIONS:
Procedure: Trans-incisional rectus sheath block — After removal of the gallbladder, a predetermined volume of 0.2% ropivacaine (1cc/kg, max dose 10cc, divided into equal doses bilaterally) will be administered under direct visualization into the rectus sheath bilaterally by the attending surgeon. This will be done after closure of the fascial incision but prior to closure of the skin incision.
  Arms: Trans-incisional rectus sheath block
Procedure: Laparoscopic guided rectus sheath block — After removal of the gallbladder, a predetermined volume of 0.2% ropivacaine (1cc/kg, max dose 10cc, divided into equal doses bilaterally) will be administered intra-abdominally under direct laparoscopic visualization into the rectus sheath bilaterally by the attending surgeon.
  Arms: Laparoscopic guided rectus sheath block
Drug: Ropivacaine — Ropivacaine is a long-acting local anesthetic. It has been shown to be effective for peripheral nerve, caudal, and lumbar/thoracic epidural blocks and produce less motor blockade than bupivacaine after caudal administration. It will be the local anesthetic used to perform the rectus sheath block for both arms.
  Other Names: Naropin

SUMMARY:
This is a prospective, double-blinded, randomized controlled study comparing the efficacy of trans-incisional rectus sheath block to laparoscopic guided rectus sheath block for pediatric single-incision laparoscopic cholecystectomy (SILC). umbilical hernia repair in children.

Patients aged 10-21 years old undergoing SILC for cholelithiasis, cholecystitis, or biliary dyskinesia will be screened for study inclusion. Eligible patients and their parents/guardians will be approached and, if agreeable, consented for the study pre-operatively. Patients will be randomized to receive either trans-incisional rectus sheath block or intra-operative rectus sheath block under direct laparoscopic visualization. Both will be done by the attending pediatric surgeon. The patient, patient guardians, select research team members, and Post anesthesia care unit (PACU) staff will be blinded to the method of analgesic administration.

DETAILED DESCRIPTION:
Regional anesthesia has been increasingly utilized for providing post-operative analgesia for a number of surgical procedures in children. Rectus sheath block and local anesthetic infiltration of the surgical site are two common modes for providing post-operative analgesia. Studies comparing the two modes have shown ultrasound-guided rectus sheath block to improve immediate pain scores and reduce use of post-operative analgesia in pediatric patients undergoing umbilical hernia repair. However, these studies have compared pre-incisional ultrasound-guided rectus sheath block to post-operative local anesthetic infiltration as a subcutaneous and/or intradermal injection. Also, to our knowledge, there are no studies evaluating the use or efficacy of laparoscopic guided rectus sheath block for pediatric single-incision laparoscopic surgery. Single-incision surgery involves performing abdominal operations though a single, small incision, usually located at the umbilicus.

The purpose of this study is to compare the efficacy of trans-incisional rectus sheath block to intra-operative infiltration of the rectus sheath under direct laparoscopic visualization via an intra-abdominal approach for providing post-operative analgesia following single-incision laparoscopic cholecystectomy (SILC) in children.

The investigators propose a prospective study where pediatric patients who are undergoing single-incision laparoscopic cholecystectomy will be randomized pre-operatively to receive either a trans-incisional rectus sheath block after facial closure but prior to skin closure or intra-operative infiltration of the rectus sheath under direct laparoscopic visualization after cholecystectomy. The primary outcome is the post-operative pain rating based on the Wong-Baker Faces Pain Rating Scale (WBFPRS) following SILC. Additional outcomes measured will include: operative times, the use of intravenous/oral opioid and/or non-opioid medication in the post-operative period, duration of analgesia following surgery based on time to first rescue analgesic, intra-operative hemodynamic changes, post-operative hemodynamic changes, incidence of side-effects, and complications. Patients/patient guardians will receive a sheet to document post-operative WBFPRS scores, oral opioid and non-opioid medication administration once discharged to home for a total of 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 10-21 years old undergoing single-incision laparoscopic cholecystectomy

Exclusion Criteria:

* Patients with choledocolithiasis, gallstone pancreatitis, or sickle cell disease
* Allergy to bupivacaine
* Concurrent surgical procedure
* Developmental delay or neurologic diagnosis that would interfere with post- operative pain score assessment
* Chronic pain medication use, chronic pain disorder or complex regional pain syndrome
* Anesthesiologist classification of III or greater

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2015-06; Primary Completion 2018-10-01 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M Chandler, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trans-incisional Rectus Sheath Block | Laparoscopic Guided Rectus Sheath Block
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trans-incisional Rectus Sheath Block | Laparoscopic Guided Rectus Sheath Block | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.83 (1.63) | 14.83 (4) | 15.33 (3.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Pain Rating
Description: Using the Wong-Baker FACES Pain Rating Scale (WBFPRS). The WBFPRS is a visual pain rating scale in which the participant looks at pictures of faces depicting levels of pain and chooses the one that most closely resembles their own pain. The scale ranges from 0 "no hurt" to 10 "Hurts Worst."
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trans-incisional Rectus Sheath Block | Laparoscopic Guided Rectus Sheath Block
Number analyzed (Participants) | 24 | 24
score on a scale | 4.03 (1.46) | 4.03 (1.16)

2. Secondary Outcome: Operative Time
Description: Operative time is measured as the time between X and Y. Reported in minutes.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Trans-incisional Rectus Sheath Block | Laparoscopic Guided Rectus Sheath Block
Number analyzed (Participants) | 24 | 24
minutes | 62 (27) | 60 (19)

3. Secondary Outcome: Use of Post-operative Intravenous/Oral Opioid and Non-opioid
Description: Amount of postoperative intravenous/oral opioid and non-opioid medications received by patient. This is being recorded as Morphine milligram equivalents (MME)/kilogram(kg) for days 1-5.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: MME/kg
Arm/Group | Trans-incisional Rectus Sheath Block | Laparoscopic Guided Rectus Sheath Block
Number analyzed (Participants) | 24 | 24
MME/kg | 0.49 (0.32) | 056 (.42)

4. Secondary Outcome: Time to First Rescue Analgesic
Description: Amount of time in minutes until the first analgesic is given postoperatively.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Trans-incisional Rectus Sheath Block | Laparoscopic Guided Rectus Sheath Block
Number analyzed (Participants) | 24 | 24
minutes | 14.4 (11.3) | 17.9 (16.8)

5. Secondary Outcome: Number of Participants With Side Effects
Description: Number of participants with side effects such as nausea, vomiting, allergic reactions.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Trans-incisional Rectus Sheath Block | Laparoscopic Guided Rectus Sheath Block
Number analyzed (Participants) | 24 | 24
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Complications
Description: Number of participants with complications such as infection, bleeding, intravascular injection, bowel puncture.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Trans-incisional Rectus Sheath Block | Laparoscopic Guided Rectus Sheath Block
Number analyzed (Participants) | 24 | 24
Participants | 0 | 0

7. Secondary Outcome: Total Number of Complications
Description: Total number of complications such as infection, bleeding, intravascular injection, bowel puncture.
Time Frame: 30 days
Measure: Number; unit: complications
Arm/Group | Trans-incisional Rectus Sheath Block | Laparoscopic Guided Rectus Sheath Block
Number analyzed (Participants) | 24 | 24
complications | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Trans-incisional Rectus Sheath Block | Laparoscopic Guided Rectus Sheath Block
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/24 | 1/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trans-incisional Rectus Sheath Block (N=24) | Laparoscopic Guided Rectus Sheath Block (N=24)
readmission (Hepatobiliary disorders) | 1 (1) | 0 (0) — Common bile duct stone following cholecystectomy that required Endoscopic retrograde cholangiopancreatography (ERCP)
readmission (Renal and urinary disorders) | 1 (1) | 0 (0) — urinary retention requiring urinary catheterization and hospitalization
Attempted suicide (Psychiatric disorders) | 0 (0) | 1 (1) — Attempted suicide that required hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT02494336/Prot_SAP_001.pdf